CLINICAL TRIAL: NCT05944757
Title: Compare of PRP Autologous Serum and Autologous Serum by Intrastromal Injection in Different Eye Disease Conditions
Acronym: prp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Anita Syla Lokaj (Other)
Responsible Party: Sponsor-Investigator, Anita Syla Lokaj, Principal investigator Faruk Semiz, Eye Hospital Pristina Kosovo
Organization: Eye Hospital Pristina Kosovo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Anita Syla 1983
Record Dates: First submitted 2022-02-27; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: PRP
Keywords: PRP; Dry Eye; Keratoconus; Dystrophy; Regenerative therapy
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconus

STUDY DESIGN:
Intervention Model Description: Both models participated in this study.Models aged were from 20 up to 70
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP -plasma rich platelets group (Experimental): Twenty patients (20) underwent 0.5 ml intrastromal injection of PRP plasma rich platelets (first group) every 2 weeks for one month
  Interventions: Drug: PRP plasma rich platelets
- Autologous serum group (Active Comparator): Twenty patients (20) underwent intrastromal injection of 0.5 ml of autologous serum (second group) every 2 weeks for 1 month
  Interventions: Drug: Autologous serum

INTERVENTIONS:
Drug: PRP plasma rich platelets — Twenty patients (20) underwent 0.5 ml 100 % intrastromal injection of PRP plasma rich platelets (first group) every 2 weeks for one month
  Other Names: PRP
  Arms: PRP -plasma rich platelets group
Drug: Autologous serum — Twenty patients (20) underwent intrastromal injection of 0.5 ml 100 %of autologous serum (second group) every 2 weeks for 1 month
  Other Names: AS
  Arms: Autologous serum group

SUMMARY:
Platelet-rich plasma (PRP) is an autologous blood product rich in proteins and growth factors. Its application has been the subject of many studies in the field of ophthalmology to stimulate tissue healing and regeneration. Due to its anatomical features (lack of blood vessels), the cornea is among the most susceptible to damage structures of the eye. Therefore, the study of the impact of various regenerative therapies (autologous blood products, serums, ) on corneal lesions is important not only scientifically, but also practically for ophthalmologist. Numerous reports described the healing effect of PRP on corneal lesions.

DETAILED DESCRIPTION:
Purpose The objective of the study is to compare the efficacy of 100% prp autolog serum eye drops with 100 % of intrastromal injection-rich plateles plasma autolog serum eye drops in patients with moderate to severe dry eye in keratoconus disease,corneal dystrophy,chemical burns.

Methods A total of 40 eyes were included in this prospective study. Clinical records of 20 consecutive patients with dry eye disease who had been treated with conventional autolog eye drops via intrastromal injection(conventional treatment group) and 20 consecutive patients treated with intrastromal autologous PRP eye drops i(PRP eye drops treated group) from September 2021.

ELIGIBILITY:
Inclusion Criteria:

* Dry eye diseases from other conditions( diabetes,allergy,keratoconus and others)
* Corneal dystrophy
* Chemical burns
* Keratoconus

Exclusion Criteria:

* Hemoglobin saturation (less than 11 mg/dl);
* hepatopathies;
* nephropathies;
* coagulopathies;
* hemoglobinopathies;
* decompensated heart diseases;
* infectious diseases such as Chagas, syphilis, HIV, HTLV, hepatitis B and C, and others transmissible by blood considered.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Improving dry eye symptoms | 12 months
  hange From Baseline in Ocular Surface Staining [

SECONDARY OUTCOMES:
Improving corneal transparency | 12 months
  Change From Baseline in Ocular Surface Disease Index (OSDI) The OSDI consists of 12 questions on items related to the assessment of symptoms, functional limitations and environmental factors related to dry eye. It is graded on a scale of 0-4, with 0 indicating none of the time, 1 for some of the time, 2 for half of the time, 3 for most of the time and 4 indicating all the time. This is a valid and reliable instrument for measuring the severity of dry eye.
  The total OSDI score was then calculated by the following formula: OSDI = (sum of scores for all questions answered) × 100/(total number of questions answered) × 4). A score of 0-100 was obtained, related to the extent of dry eye, which a higher score representing greater symptoms severity.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Syla Lokaj, Principal Investigator — Eye Hospital,Univeristy Center Clinic of Kosova
Locations (1):
- Eye Hospital,University Center Clinic of Kosova, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No